CLINICAL TRIAL: NCT05111041
Title: Development of a M-Health Smokeless Tobacco Cessation Intervention for Firefighters
Brief Title: Smokeless Tobacco Cessation Intervention for Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109404; 5R01CA242593-03 (NIH)
Record Dates: First submitted 2021-11-01; First posted 2021-11-08 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Smokeless Tobacco Cessation
Keywords: Firefighters; Smokeless Tobacco; Quitting Smokeless Tobacco; First Responders
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- #EnufSnuff.TXT- First Responder (Experimental): Participants in this group will receive a mobile gradual smokeless tobacco reduction intervention
  Interventions: Behavioral: #EnufSnuff.TXT- First Responder
- Enough Snuff Intervention (Active Comparator): Participants in this group will receive tobacco cessation materials
  Interventions: Behavioral: Enough Snuff Intervention

INTERVENTIONS:
Behavioral: #EnufSnuff.TXT- First Responder — Participants in this intervention will be given the choice of following the Gradual Reduction to Quit program or to choose their own quit date within 2-4 weeks. The Gradual Reduction to Quit program will reduce smokeless tobacco use via text message support and weekly prompts guiding the participants to gradually decrease their use of smokeless tobacco until they are down to zero. A four week Nicotine Replacement Therapy (NRT) sample in the form of lozenges will also be provided to all participants. The intent of this program is to reduce the number of times participants use smokeless tobacco.
  Arms: #EnufSnuff.TXT- First Responder
Behavioral: Enough Snuff Intervention — Participants will be sent the Enuf Snuff cessation manual, support text messages, as well as a four week Nicotine Replacement Therapy (NRT) sample in the form of lozenges.
  Arms: Enough Snuff Intervention

SUMMARY:
The investigators are asking professional firefighters across North Carolina to take part in focus groups to discuss the specific needs of firefighters in smokeless tobacco cessation. About 40 firefighters will take part in the focus groups.

The purpose of the focus groups is to learn how firefighting and shift work impact smokeless tobacco use and risk perceptions related to chew or dip. Using their feedback, the study team will then develop a cessation program specifically geared towards firefighters and first responders.

The cessation program will be a mobile text / chat intervention specifically tailored to needs of firefighters and first responders who wish to stop using smokeless tobacco. About 50 firefighters and first responders will take part in this program, while being randomized into either the intervention group or the control group.

ELIGIBILITY:
Inclusion Criteria:

* Professional firefighters or first responders
* 18 years or older
* Have used smokeless tobacco for the past year and current (past 30 days) smokeless tobacco daily use
* Access to a smartphone

Exclusion Criteria:

* Not a professional firefighter or first responder
* Under 18 years of age
* Have not used smokeless tobacco for the past year and are not current (past 30 days) smokeless tobacco daily use
* No access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noonan D, Fish LJ, Silva SG, Da Costa M, Simmons LA, Garcia Ortiz N, Swinkels C, Jung D, Severson HH, Pollak KI. #EnufSnuff.TXT-FirstResponder: a pilot randomized controlled trial of a text message intervention for smokeless tobacco cessation among First Responders. Front Public Health. 2026 Jan 19;13:1699800. doi: 10.3389/fpubh.2025.1699800. eCollection 2025. PMID 41635441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited using social media (i.e., Facebook). An advertising profile for the study targeted the study population (e.g., current smokeless tobacco users (chewer/dipper), at or over age 18, currently working or volunteering as a firefighter or first responder, with access to a smartphone). This was a single-site study, which used electronic consents and survey measures.
Pre-assignment Details: Participants were required to verify their age, location, and smokeless tobacco use when submitting their information via the advertisement. During the electronic screener survey, participants were required to verify their age, first responder status, and use of smokeless tobacco as well. If any answers were outside of the eligibility requirements, they were directed to an ineligibility notification screen in the RedCap system. Those deemed eligible proceeded to the Baseline survey.
Groups:
- #EnufSnuff.TXT- First Responder: Participants in this group will receive a mobile gradual smokeless tobacco reduction intervention and support text messages.
  #EnufSnuff.TXT- First Responder: Participants in this intervention will be given the choice of following the Gradual Reduction to Quit program or to choose their own quit date within 2-4 weeks. The Gradual Reduction to Quit program will reduce smokeless tobacco use via text message support and weekly prompts guiding the participants to gradually decrease their use of smokeless tobacco until they are down to zero. A four week Nicotine Replacement Therapy (NRT) sample in the form of lozenges will also be provided to all participants. The intent of this program is to reduce the number of times participants use smokeless tobacco.
- Enough Snuff Intervention: Participants in this group will receive tobacco cessation materials and support text messages.
  Enough Snuff Intervention: Participants will be sent the Enuf Snuff cessation manual, support text messages, as well as a four week Nicotine Replacement Therapy (NRT) sample in the form of lozenges.
Period: Overall Study
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Started | 30 | 30
Completed | 23 | 23
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 6 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (9.6) | 37.7 (10.4) | 37.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of First Responders Recruited Who Completed a Screening Assessment
Time Frame: Within 3 months of the initiation of study recruitment
Population: First responders recruited and screened for the study.
Measure: Count of Participants; unit: Participants
Groups:
- Recruited First Responders: First responders recruited and screened for the study.
Arm/Group | Recruited First Responders
Number analyzed (Participants) | 163
Participants | 163

2. Primary Outcome: First Responders Who Met the Study Eligibility Criteria, Were Enrolled, and Randomized to a Treatment Arm
Time Frame: Within 3 months of the initiation of study recruitment
Population: First responders who met the study eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

3. Primary Outcome: Percent of Participants Engaged With the Program as Measured by Completion of the End of Program Questionnaire
Description: Study engagement defined as completing the End of Intervention Program assessment.
Time Frame: 30 days following the end of the 10-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 23 | 23
Statistical Analysis 1: Comparison: #EnufSnuff.TXT- First Responder vs Enough Snuff Intervention; Test type: Superiority; p = 1.000, Regression, Logistic — Not adjusted for multiple outcomes due to exploratory nature of the study; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.302 to 3.309]

4. Primary Outcome: Number of Participants Who Stated Intervention Was Useful as Measured by Questionnaire
Description: Usefulness was measured on a scale of 1-5, where 1=Not at all useful, 2=Somewhat useful, 3=Undecided, 4=Very useful, 5=Extremely useful. Ratings were dichotomized for the analysis as 0=no (not at all, somewhat, undecided) or 1=yes (very, extremely useful).
Time Frame: 30 days following the end of the 10-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 5 | 6
Statistical Analysis 1: Comparison: #EnufSnuff.TXT- First Responder vs Enough Snuff Intervention; Test type: Superiority; p = 0.7389, Regression, Logistic — Not adjusted for multiple outcomes due to exploratory nature of the study; Odds Ratio (OR) = 0.800, 95% CI 2-sided [0.215 to 2.972]

5. Primary Outcome: Number of Participants Who Stated That #EnufSnuff.TXT Intervention Was Helpful as Measured by Questionnaire
Description: Helpfulness was measured on a scale of 1-5 where 1=not at all, 2=somewhat, 3=Undecided, 4=very, 5=extremely. Ratings were dichotomized for the analysis as 0=no (not at all, somewhat, undecided) and 1=yes (very, extremely).
Time Frame: 30 days following the end of the 10-week intervention
Population: Not relevant to the Enough Snuff Intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 0
Participants | 9 |

6. Primary Outcome: Number of Participants Who Stated Intervention Made Them Consider Quitting as Measured by Questionnaire
Description: Considered quitting was measured on a scale of 1-5, where 1=Not at all useful, 2=Somewhat useful, 3=Undecided, 4=Very useful, 5=Extremely useful. Ratings were dichotomized for the analysis as 0=no (not at all, somewhat, undecided) or 1=yes (very, extremely useful).
Time Frame: 30 days following the end of the 10-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 16 | 14
Statistical Analysis 1: Comparison: #EnufSnuff.TXT- First Responder vs Enough Snuff Intervention; Test type: Superiority; p = 0.6058, Regression, Logistic — Not adjusted for multiple outcomes due to exploratory nature of the study; Odds Ratio (OR) = 1.306, 95% CI 2-sided [0.474 to 3.602]

7. Primary Outcome: Number of Participants Who Stated They Would Recommend Program to a Friend as Measured by Questionnaire
Description: Recommend to friend was measured on a scale of 1-5, where 1=Not at all useful, 2=Somewhat useful, 3=Undecided, 4=Very useful, 5=Extremely useful. Ratings were then dichotomized for the analysis as 0=no (not at all, somewhat, undecided) or 1=yes (very, extremely useful).
Time Frame: 30 days following the end of the 10-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 11 | 11
Statistical Analysis 1: Comparison: #EnufSnuff.TXT- First Responder vs Enough Snuff Intervention; Test type: Superiority; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.349 to 2.866]

8. Primary Outcome: Number of Participants Who Quit Smokeless Tobacco Measured by Self Report
Description: Quit was determined by the self-report response (yes or no) to the question, "In the past 7 days, have you used any dip?"
Time Frame: 30 days following the end of the 10-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
Number analyzed (Participants) | 30 | 30
Participants | 12 | 10
Statistical Analysis 1: Comparison: #EnufSnuff.TXT- First Responder vs Enough Snuff Intervention; Test type: Superiority; p = 0.5925, Regression, Logistic — Not adjusted for multiple outcomes due to exploratory nature of the study; Odds Ratio (OR) = 1.333, 95% CI 2-sided [0.465 to 3.823]

ADVERSE EVENTS:
Time Frame: Up to 30 days following the end of the 10-week intervention
Arm/Group | #EnufSnuff.TXT- First Responder | Enough Snuff Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT05111041/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT05111041/ICF_000.pdf